CLINICAL TRIAL: NCT01726309
Title: Correlation of Single Nucleotide Polymorphism (SNP) Profile of Domain III of EGFR to Skin Toxicity and Disease Response to Treatment With Erbitux Requirements
Brief Title: Single Nucleotide Polymorphism(SNP)Study. ICORG 08-40, V4
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 08-40
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Stage IV CRC
- Stage IV NSCLC

SUMMARY:
Primary Objective:

Correlation of the skin and/or eye toxicity grade secondary to Cetuximab or Panitumumab and the SNP profile of the Epidermal Growth Factor Receptor (EGFR) domain III region.

Secondary Objectives:

Correlation of SNP profile with indicators of tumour response parameters, such as radiological response, duration of response, time to progression (TTP), overall survival (OS) time, incidence of non-dermatological adverse events.

DETAILED DESCRIPTION:
Baseline assessment:

* Contact Lenses
* Medical History
* Previous chemotherapy
* Vital Signs (weight, height, Karnofsky Performance status, heart rate, blood pressure)
* Symptom Assessment (Pre-existing skin and/or eye conditions, CEA measurement (CRC only), Disease status (TNM Staging))
* Planned chemotherapy regimen
* Radiotherapy

Blood Sample: A 2ml blood sample should be collected in ethylenediamine-tetraacetic acid (EDTA) containing Vacutainer at any time before or after starting treatment. DNA will be extracted from the samples and the 11 SNPs in the region of the EGFR gene encoding domain III will be characterized.

Follow-up Assessment: with every second cycle of Cetuximab- or Panitumumab-containing regimen (CRC: every 2. Week; NSCLC: every 3-4 weeks):

* Visit Number and Date
* Vital Signs (weight, height, Karnofsky Performance status, heart rate, blood pressure)
* Symptom Assessment (CEA measurement (CRC only), Disease status (TMN Staging), Skin Toxicity (CTCAE) grading)
* Current chemotherapy regimen
* Radiotherapy
* CEA measurement only for CRC (every second cycle/every 4 weeks)

Long-term follow-up (up to 5 years):

* CT restaging (TNM Staging) should be done 3 monthly for as long as the subject is receiving Cetuximab- or Panitumumab- containing regimen or if there is suspicion of disease progression.
* OS

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV (AJCC 7th Edition TMN Staging, Appendix C), histologically confirmed CRC with wild-type KRAS and not a candidate for metastasectomy.
2. Stage IV (AJCC 7th Edition, TMN Staging, Appendix C) NSCLC expressing EGFR (IHC tested)
3. Patients, who will receive treatment with an EGFR-antibody (Cetuximab or Panitumumab).
4. Karnofsky performance status (Appendix B) score ≥60.
5. Acceptable laboratory values:

   * Haemoglobin ≥ 9 g/dL.
   * Neutrophil count ≥ 1.0 x 10^9/L.
   * Platelet count ≥100 x 10^9/L.
   * Serum creatinine ≤1.5 times the upper limit of normal.
   * Bilirubin ≤1.5 times the upper limit of normal.
   * Aspartate aminotransferase and alanine aminotransferase ≤5 times the upper limit of normal.

Exclusion Criteria:

1. Aged < 18 years
2. Prior exposure to Cetuximab or Panitumumab
3. The CRC does not carry wild-type KRAS.
4. The NSCLC stains negative for EGFR protein expression
5. Second cancer diagnosis (apart from non-melanoma skin cancer)
6. Known hypersensitivity to Cetuximab or Panitumumab, or murine protein.
7. Known history of coronary artery disease, arrhythmias, or congestive heart failure (If the treating physician feels that a patient's coronary artery disease / arrhythmia / congestive heart failure does not place him/her at risk from treatment with an anti-EGFR antibody, the person can be included. This is a clinical decision, which has to be made by the treating physician).
8. Known to be pregnant (pregnancy test is not mandatory) or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Population:
  150 Patients with histologically proven stage IV (AJCC 7th Edition) colorectal cancer (CRC) expressing wild-type KRAS or stage IV non-small cell lung cancer (NSCLC) expressing EGFR (tested by immunohistochemistry (IHC)), with no previous exposure to Cetuximab or Panitumumab, who will receive treatment with an EGFR-antibody (Cetuximab or Panitumumab).
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Correlation between the type and degree of reported skin and/or eye reaction and the SNP profile of the EGFR domain III region. | Throughout treatment with up to 5 years in follow up
  Using Common Terminology Criteria for Adverse Events (CTCAE) version 4

SECONDARY OUTCOMES:
Correlation between the SNP profile(s) and disease response | Throughout treatment with up to 5 years in follow up
  Time to progression TTP and OS over 5 years

CONTACTS AND LOCATIONS:
Locations (10):
- Ireland (10):
  - Letterkenny General Hospital, Letterkenny, Donegal
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - The Adelaide & Meath Hosptal, Dublin Incorporating The National Children's Hospital, Dublin
  - Galway University Hospital, Galway
  - Our Lady of Lourdes Hospital, Drogheda, Louth
  - Waterford Regional Hospital, Waterford